CLINICAL TRIAL: NCT00409708
Title: An Open-label, Behavioral-treatment-controlled Evaluation of the Effects of Extended Release Methylphenidate on the Frequency of Cytogenetic Abnormalities in Children 6 - 12 Years of Age With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Effects of Methylphenidate on Cellular Abnormalities in Children With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRIT124D2201
Record Dates: First submitted 2006-12-08; First posted 2006-12-11 (Estimated); Results first posted 2011-05-17 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder,; ADHD; Cytogenetic abnormalities,; extended-release methylphenidate,
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Chromosome Aberrations | interventions — Methylphenidate; Behavior Therapy

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Extended Release Methylphenidate (Ritalin LA ) plus Behavior Therapy
- 2 (Other)
  Interventions: Behavioral: Behavior Therapy

INTERVENTIONS:
Drug: Extended Release Methylphenidate (Ritalin LA ) plus Behavior Therapy
  Other Names: Ritalin LA
  Arms: 1
Behavioral: Behavior Therapy
  Arms: 2

SUMMARY:
This study will assess the frequency of chromosomal abnormalities measured in circulating lymphocytes in treatment-naive children with Attention Deficit Hyperactivity Disorder (ADHD) treated for 3 months with either extended release methylphenidate or behavioral therapy.

DETAILED DESCRIPTION:
This study will determine whether the administration of extended-release methylphenidate in treatment-naïve children with Attention Deficit Hyperactivity Disorder (ADHD) affects the frequency of chromosomal abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Children of both genders, 6-12 years old
* Written informed consent by the parent and the patient (over 7)
* Diagnosis of ADHD
* Age-appropriate cognitive functioning
* All patients who had at least one post-baseline cytogenetic assessment in the core study can enter the observation phase.

Exclusion Criteria:

* History of malignant neoplasm
* History of seizures (except childhood febrile seizures)
* Hyperthyroidism
* Concurrent medical condition which may interfere with study

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 142 (Actual)
Dates: Start 2006-11; Primary Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals Investigational site, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ritalin LA Plus Behavior Therapy: 10-60 mg/day
- Behavior Therapy: 0 mg/day Ritalin LA
Period: Treatment
Arm/Group | Ritalin LA Plus Behavior Therapy | Behavior Therapy
Started | 53 (A total of 142 participants were screened for the study but only 109 were randomized to treatment) | 56
Completed | 38 | 39
Not Completed | 15 | 17
Not completed — Abnormal test procedure result(s) | 1 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Protocol Violation | 6 | 2
Not completed — Withdrawal by Subject | 3 | 8
Not completed — Lost to Follow-up | 0 | 6
Not completed — Administrative problems | 5 | 0
Period: Washout
Arm/Group | Ritalin LA Plus Behavior Therapy | Behavior Therapy
Started | 38 | 39
Completed | 17 | 29
Not Completed | 21 | 10
Not completed — Lack of Efficacy | 9 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 11 | 5
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ritalin LA Plus Behavior Therapy | Behavior Therapy | Total
Number analyzed (Participants) | 52 | 52 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 52 | 52 | 104
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 8.3 (1.75) | 8.5 (1.91) | 8.4 (1.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 17 | 38
  Male | 31 | 35 | 66

OUTCOME MEASURES:

1. Primary Outcome: The Number of Chromosomal Aberrations Per 100 Cells Excluding Gaps at Baseline and at the End of Treatment i.e Day 84 (Week 12)
Description: The number of chromosomal aberrations per 100 cells excluding gaps at Baseline (n=33, n=32) and at Week 12 (n=33, n=32) was counted in blood samples cultured for 48 hours using a standard protocol. The types of abnormalities included translocations (reciprocal and non-reciprocal), insertions, dicentrics, fragments, inversions, chromatid exchanges (quadriradials and triradials), breaks, and other unusual observations, eg, aneuploidy, tetraploidy or endoreduplication.
Time Frame: baseline and at end of treatment (Week 12)
Population: Per-Protocol-1 (PP1) population: The PP1 population consisted of all patients who were randomized and provided cytogenetic data for at least one of the primary endpoints at baseline and at the Week 12 evaluation.
Measure: Mean (Standard Deviation); unit: number of abnormalities
Arm/Group | Ritalin LA Plus Behavior Therapy | Behavior Therapy
Number analyzed (Participants) | 36 | 35
number of abnormalities
  Baseline | 1.05 (1.246) | 0.75 (1.008)
  At the end of treatment i.e. week12: Mean | 0.53 (1.132) | 0.41 (0.665)

2. Secondary Outcome: Number of Sister Chromatoid Exchanges Per Cell
Description: Blood collected at baseline (n=20, n=14) and at the end of treatment, Week 12, (n= 20, n= 14) was cultured for 48 hours using a standard protocol. Giemsa staining and/or fluorescent in situ hybridization (FISH) chromosome painting was done on the cells in metaphase and the number of chromatoid exchanges per cell was recorded by blinded raters.
Time Frame: baseline and at end of treatment (Week 12)
Population: Per-Protocol-2 population: The PP2 population consisted of all subjects who were randomized and provided at least one post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: number of sister chromatoid exchanges
Arm/Group | Ritalin LA Plus Behavior Therapy | Behavior Therapy
Number analyzed (Participants) | 38 | 37
number of sister chromatoid exchanges
  Baseline | 7.807 (0.9228) | 7.533 (1.2160)
  At the end of treatment i.e. Week12 | 7.213 (1.0408) | 7.303 (0.6165)

3. Secondary Outcome: Pharmacokinetic/Pharmacodynamic Relationship of Methylphenidate Blood Levels and Cytogenetic Changes
Description: Since no cytogenetic effects were observed, blood samples were not analyzed for pharmacokinetics/pharmacodynamics.
Time Frame: End of treatment (Week 12)
Measure: Number; unit: Number
Arm/Group | Ritalin LA Plus Behavior Therapy | Behavior Therapy
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Baseline to End of Treatment (Week 12) on the Conners' ADHD/DSM-IV Scale for Parents (CADS-P)
Description: Parents completed the Conners' ADHD/DSM-IV Scale for Parents (CADS-P) consisting of the ADHD Index (12 items) and the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV)( 18 items). Parents rated their child's behavior of the previous week from a list of common problems. When asked "How much of a problem has this been in the last week?" parents selected 0 = none, not at all, seldom, or very infrequently; 3 = very much true, or it occurs very often or frequently; or 1 or 2 for ratings in between. A score of 50 is considered normal and more than 70 markedly atypical.
Time Frame: Baseline to end of treatment (Week 12)
Population: Per-Protocol-2 (PP2) Population: The PP2 population consisted of all subjects who were randomized and provided at least one post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Units on a rating scale
Arm/Group | Ritalin LA Plus Behavior Therapy | Behavior Therapy
Number analyzed (Participants) | 38 | 37
Units on a rating scale | -17.0 (11.23) | -7.0 (9.97)

5. Secondary Outcome: Change From Baseline to the End of Treatment (Week 12) on the Global Improvement Rating of the Clinical Global Impression Scale (CGI-I)
Description: The Clinical Global Impression scale (CGI-I) is a clinician-rated instrument designed to assess the overall change of illness relative to baseline. The CGI-I consists of 7 ratings as follows: 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. CGI-I assessments are relative to the patient's status at the Baseline visit.
Time Frame: From baseline to the end of treatment (Week 12)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a rating scale
Arm/Group | Ritalin LA Plus Behavior Therapy | Behavior Therapy
Number analyzed (Participants) | 38 | 37
Units on a rating scale | 1.9 (0.81) | 3.0 (0.97)

6. Secondary Outcome: Change From Baseline to the End of Treatment (Week 12) on the Severity of Illness Rating of the Clinical Global Impression Scale (CGI-S)
Description: The Clinical Global Impression scale (CGI-S) is a clinician-rated instrument designed to assess the severity of illness. The CGI-S rating indicates illness severity at each time-point on a scale as follows: 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = extremely ill. CGI-S assessments are relative to the patient's status at the Baseline visit.
Time Frame: From baseline to the end of treatment (Week 12)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a rating scale
Arm/Group | Ritalin LA Plus Behavior Therapy | Behavior Therapy
Number analyzed (Participants) | 38 | 37
Units on a rating scale | -1.9 (0.98) | -0.6 (1.01)

7. Primary Outcome: The Number of Micronuclei Per 1000 Binucleated Cells Endpoints at Baseline and at the End of Treatment i.e Day 84 (Week 12)
Description: The number of micronuclei per 1000 binucleated cells was measured at Baseline ( n=34 , n=29 ) and at the end of treatment, Week 12 (n =34, n= 29), in blood cultured for 48 hours using a standard protocol.
Time Frame: baseline and at end of treatment (Week 12)
Measure: Mean (Standard Deviation); unit: number of micronuclei per 1000 binucleat
Arm/Group | Ritalin LA Plus Behavior Therapy | Behavior Therapy
Number analyzed (Participants) | 36 | 35
number of micronuclei per 1000 binucleat
  At Baseline | 5.76 (2.336) | 5.71 (4.535)
  At the end of treatment i.e. Week 12 | 3.63 (2.053) | 4.19 (2.737)

ADVERSE EVENTS:
Groups:
- Ritalin+Behavior: Ritalin+Behavior
- Behavior: Behavior
Arm/Group | Ritalin+Behavior | Behavior
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 28/52 | 13/52
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ritalin+Behavior (N=52) | Behavior (N=52)
Abdominal Pain Upper (Gastrointestinal disorders) | 5 | 2
Vomiting (Gastrointestinal disorders) | 5 | 1
Fatigue (General disorders) | 4 | 0
Pyrexia (General disorders) | 2 | 3
Nasopharyngitis (Infections and infestations) | 4 | 4
Upper Respiratory Tract Infection (Infections and infestations) | 6 | 5
Decreased Appetite (Metabolism and nutrition disorders) | 10 | 0
Headache (Nervous system disorders) | 7 | 1
Initial Insomnia (Psychiatric disorders) | 3 | 0
Insomnia (Psychiatric disorders) | 5 | 0
Tearfulness (Psychiatric disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1

LIMITATIONS AND CAVEATS:
Since no cytogenetic effects were observed, blood samples were not analyzed for pharmacokinetics/pharmacodynamics.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.